CLINICAL TRIAL: NCT00073502
Title: A Phase II Study of Single Agent OSI-7904L In Patients With Locally Advanced or Metastatic Adenocarcinoma Of the Stomach or Gastroesophageal Junction
Brief Title: Phase II Study of Single Agent OSI-7904L in Patients With Gastric or Gastroesophageal (GEJ) Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: OSI Pharmaceuticals (Industry)
Purpose: Treatment
Other Study IDs: OSI-904-201
Record Dates: First submitted 2003-11-21; First posted 2003-11-25 (Estimated); Last update posted 2006-02-22 (Estimated); Status verified 2003-10

CONDITIONS: Gastroesophageal Adenocarcinoma; Gastric Adenocarcinoma
MeSH Terms: interventions — ((S)-2-(5-(1,2-dihydro-3-methyl-1-oxobenzo(f)-quinazoline-9-yl)methyl)amino-1-oxo-2-isoindolynyl)-glutaric acid

INTERVENTIONS:
Drug: OSI-7904L

SUMMARY:
Multi-center, open-label, non-randomized Phase II study to evaluate the efficacy and safety of OSI-7904L in gastric and GEJ cancers. Those patients who do not derive clinical benefit after two cycles may be switched to a commonly used combination regimen.

ELIGIBILITY:
Inclusion Criteria:

Documented locally advanced or metastatic adenocarcinoma of the stomach or gastroesophageal junction No prior chemotherapy for locally advanced or metastatic disease Adequate baseline bone marrow, hepatic and renal function Age >= 18 years At least one target lesion

Exclusion Criteria:

Active or uncontrolled infections or other serious illnesses or other medical conditions (eg, hepatitis, HIV, chronic alcohol abuse) Symptomatic brain metastases which are not stable

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43
Dates: Start 2003-10; Study Completion 2003-10

CONTACTS AND LOCATIONS:
Locations (11):
- United States (3):
  - University of Pennsylvania Cancer Center, Philadelphia, Pennsylvania
  - MD Anderson Cancer Center, Houston, Texas
  - University of Utah, Huntsman Cancer Institute, Salt Lake City, Utah
- Dept Internal Medicine Gastrointestinal Oncology Unit, B-3000 Leuven, Belgium
- United Kingdom (7):
  - Bristol Haematology & Oncology Centre, Bristol, Avon
  - ICRF Medical Oncology Unit, Oxford, Oxfordshire
  - Deanesly Centre, Wolverhampton, West Midlands
  - NICCTU, East Podium, C-Floor, Belfast
  - Beatson Oncology Centre, Glasgow
  - Cookridge Hospital, Leeds
  - Department of Medical Oncology, Manchester